CLINICAL TRIAL: NCT04093102
Title: Role of Biomarkers to Screen for Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Abuzaid Ali, Principal Investigator, Assiut University
Other Study IDs: obstructive sleep apnea
Record Dates: First submitted 2019-08-12; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Environmental Biomarkers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: cases with obsrtuctive sleep apnea
  Interventions: Diagnostic Test: biomarkers
- control: cases without obstructive sleep apnea.
  Interventions: Diagnostic Test: biomarkers

INTERVENTIONS:
Diagnostic Test: biomarkers — bio-markers testing will be made to all suspected OSA patients(CRP, Hba1C,uric acid, ESR, plasma fibrinogen, pentraxin3), and to control cases.

SUMMARY:
assess the relationship between obstructive sleep apnea and endocrine, inflammatory, and metabolic bio-markers in consecutively enrolled adult male patients with a clinical suspicion of obstructive sleep apnea.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a disorder with high prevalence, estimated to occur in 34% of men and 17% of women , afflicting more than 100 million adults worldwide.

OSA is the third most common serious respiratory condition after Asthma and COPD.

Patients with untreated OSA are at increased risk for hypertension, cardiovascular disease, heart failure, stroke, obesity, metabolic dysregulation, diabetes mellitus, daytime sleepiness, depression, accidents and are a significant burden on the healthcare system.

Unfortunately, up to 90% of individuals with OSA remain without a diagnosis or therapy.

The association between OSA and adverse health consequences has led the American Heart Association and others to suggest that OSA screening be integrated into routine clinical care.

Current tools for OSA screening rely on questionnaires with low diagnostic accuracy from low-quality studies, as reported in meta-analyses, OSA screening measures that are frequently used include the Epworth Sleepiness Scale (ESS) and STOP-Bang questionnaires.

The ESS assesses subjective daytime sleepiness but is nonspecific for OSA, was not designed nor validated for OSA screening.

The recent American Academy of Sleep Medicine (AASM) clinical practice guidelines report that more accurate and user-friendly screening tools, such as blood bio-markers, are needed to better predict OSA diagnosis and severity, a recent review of potential OSA bio-markers concludes that an optimal screening test should be clinically sensitive, specific, simple, timely, inexpensive, and correlate to disease severity.

Furthermore, bio-markers should make pathophysiological sense, reflecting functional changes that accompany OSA.

Numerous individual OSA blood bio-markers have been studied previously dysfunctions in metabolic and endocrine systems induced by OSA, chronic inflammation, hypoxemia, sleep fragmentation, and stress are associated with alterations in bio-markers. These bio-markers include glycated hemoglobin (HbA1c), C-reactive protein (CRP), erythropoietin (EPO), and uric acid,Unfortunately, the diagnostic utility of individual bio-markers or combinations of markers is inconclusive in identifying OSA.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a clinical suspicion of obstructive sleep apnea enrolled to the investigator's chest department.

Exclusion Criteria:

* Patients who previously treated as obstructive sleep apnea, or receiving opioid pain medications.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: it will be patients with suspected OSA , bio-markers testing and polysomnography will be done for all participants.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Validity of biomarkers to screen for obstructive sleep apnea | baseline
  analysis of biomarkers results (which include Pentraxin 3, HbA1C,Uric acid,CRP,ESR,Plasma fibrinogen) will be assessed and compared to the results of polysymnography

SECONDARY OUTCOMES:
Inflammatory biomarker level in OSA patients compared to controls | baseline
  Inflammatory biomarkers which include ESR , CRP and pentraxin 3 will be measured and compared in both cases and controls.

CONTACTS AND LOCATIONS:
Overall Officials: suzan salama, professor, Study Director

REFERENCES:
- [Background] Watson NF. Health Care Savings: The Economic Value of Diagnostic and Therapeutic Care for Obstructive Sleep Apnea. J Clin Sleep Med. 2016 Aug 15;12(8):1075-7. doi: 10.5664/jcsm.6034. PMID 27448424
- [Background] Kapur V, Blough DK, Sandblom RE, Hert R, de Maine JB, Sullivan SD, Psaty BM. The medical cost of undiagnosed sleep apnea. Sleep. 1999 Sep 15;22(6):749-55. doi: 10.1093/sleep/22.6.749. PMID 10505820
- [Background] Maeder MT, Mueller C, Schoch OD, Ammann P, Rickli H. Biomarkers of cardiovascular stress in obstructive sleep apnea. Clin Chim Acta. 2016 Sep 1;460:152-63. doi: 10.1016/j.cca.2016.06.046. Epub 2016 Jul 2. PMID 27380998
- [Background] Montesi SB, Bajwa EK, Malhotra A. Biomarkers of sleep apnea. Chest. 2012 Jul;142(1):239-245. doi: 10.1378/chest.11-2322. PMID 22796846